CLINICAL TRIAL: NCT01855997
Title: A Phase IV, Blood Sample Collection Study For Exploratory Evaluation of the Association of Single Nucleotide Polymorphisms With Treatment Responses From Subjects With HBe-Antigen Positive or Negative Chronic Hepatitis B, Who Received Therapy for Hepatitis B With Peginterferon Alfa-2a 40kD (Peg-IFN) ± Nucleos(t)Ide Analogue
Brief Title: A Study to Collect Blood Biomarker Samples From Participants With Chronic Hepatitis B (CHB) Who Received Treatment With Pegasys (Peginterferon Alfa-2a) ± Nucleoside/Nucleotide Analogue
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: GV28855
Record Dates: First submitted 2013-05-08; First posted 2013-05-17 (Estimated); Results first posted 2016-04-08 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood samples

GROUPS / COHORTS (1):
- Adult CHB Participants Treated With Peg-IFN Alfa-2a: Adult participants with CHB infection, and who have completed at least 24 weeks of Peg-IFN alfa-2a with/without nucleoside analogue therapy and at least 24 weeks of follow-up, will be included. Participants will be recruited from Roche clinical trials or general practice; no treatment will be administered in this non-interventional study.
  Interventions: Drug: Peg-IFN alfa-2a

INTERVENTIONS:
Drug: Peg-IFN alfa-2a — Participants received Peg-IFN alfa-2a prior to enrollment for at least 24 weeks. Dosing was chosen according to standard of care or at the discretion of the treating physician.
  Other Names: Pegasys

SUMMARY:
This Phase 4 study is designed for the collection of blood biomarker samples from participants who have completed CHB treatment with at least 24 weeks of a pegylated interferon alfa-2a (Peg-IFN alfa-2a) containing regimen and at least 24 weeks post-treatment follow-up. Participants may be enrolled from historical studies supported or sponsored by Roche, ongoing studies supported or sponsored by Roche, or from general medical practice. The follow-up of individuals who choose to participate in this study will be in accordance with the ongoing studies or with the general medical practice of the physician. Data from whole blood deoxyribonucleic acid (DNA) samples collected in the GV28555 study or available from previously collected Roche Clinical Repository (RCR) samples will be used for combined analysis with data from other applicable studies. Procedures will include blood sample collection (not applicable for participants who previously have consented and donated RCR DNA samples) and medical record capture.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to (≥) 18 years of age
* CHB
* Previously enrolled in a Roche study and treated for CHB for ≥24 weeks with Peg-IFN ± nucleoside analogue (lamivudine or entecavir) or Peg-IFN ± nucleotide analogue (adefovir) and with ≥24 weeks post-treatment follow-up; or
* Treated in general practice for CHB with Peg-IFN according to standard of care and in line with the current Summary of Product Characteristics (SmPC)/local labeling who have no contraindication to Peg-IFN therapy as per local label and have been treated with Peg-IFN for ≥24 weeks and have ≥24 week post-treatment response available at the time of blood sample collection

Exclusion Criteria:

* Hepatitis A, hepatitis C, or human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CHB who received therapy with Peg-IFN ± nucleoside/nucleotide analogue will be included.
Sampling Method: Probability Sample
Enrollment: 1669 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2014-11-28 (Actual); Study Completion 2014-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (84):
- Medizinische Universität Wien; Univ.Klinik für Innere Medizin III - Gastroenterologie & Hepatologie, Vienna, Austria
- Bulgaria (2):
  - MHAT Tokuda Hospital Sofia; Department of Gastroenterology at Clinic of Internal Deseases, Sofia
  - Mhat Sveta Marina; Clinic of Gastroenterology, Varna
- China (25):
  - Beijing Ditan Hospital, Beijing
  - Beijing 302 Hospital; No. 2 Infectious Disease Section, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing You An Hospital; Digestive Dept, Beijing
  - Xiangya Hospital of Centre-South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The Second Affiliated Hospital, Chongqing Medical University, Chongqing
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The Eighth People's Hospital of Guangzhou, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - Hangzhou Sixth People's Hospital, Hangzhou
  - The 1st Affiliated Hospital of Harbin Medical University, Harbin
  - Jinan Infectious Diseases Hospital, Jinan
  - Nanjing No.2 Hospital; Liver Disease Department, Nanjing
  - The First Affiliate Hospital of Guangxi Medical University, Nanning
  - Shuguang Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - Shenzhen Donghu Hospital, Shenzhen
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - Xinjiang Uygur Autonomous Region Hospital of Chinese Traditional Medicine, Ürümqi
  - Tongji Hosp, Tongji Med. Col, Huazhong Univ. of Sci. & Tech, Wuhan
  - The Second Affiliated Hospital of The Fourth Military Medical University (Tangdu Hospital), Xi'an
  - General Hospital of Ningxia Medical University, Yinchuan
  - Henan Provincial People's Hospital, Zhengzhou
- France (4):
  - Hopital Beaujon;Hepatologie, Clichy
  - Hopital Henri Mondor; Hepatologie Gastro Enterologie, Créteil
  - Hopital de Pontchaillou; Medicine Interne - Hepatologie, Rennes
  - Institut Arnault Tzanck; Medecine I Gastro Enterologie, Saint-Laurent-du-Var
- Germany (5):
  - Praxis Dr. med. Christine John, Berlin
  - Praxis Dr. Heyne, Berlin
  - Charité Uni.-medizin Berlin, Campus Virchow-Klinikum; Med. Klinik m.S. Hepatologie Gastroenterologie, Berlin
  - Ifi- Studien und Projekte GmbH, An der Asklepios Klinik St. Georg, Hamburg
  - Medizinische Hochschule Zentrum Innere Medizin Abt.Gastroenterologie, Endokrinologie und Hepatologie, Hanover
- Greece (3):
  - Laiko General Hospital Athen; Uni Clinic of Gastrenterology, Athens
  - University Hospital of Larissa; Pathological Clinic, Larissa
  - Hippokratio Hospital; 4Th Internal Medicine Dpt, Thessaloniki
- Italy (12):
  - Azienda Ospedaliera Policlinico Consorziale di Bari; Clinica Malattie Infettive, Bari, Apulia
  - Ospedale de Bellis; Reparto Medicina Generale, Castellana Grotte, Apulia
  - Az. Osp. S. Sebastiano; Divisione Malattie Infettive, Caserta, Campania
  - Az. Osp. Cardarelli; Unita Operativa A Struttura Complessa Di Epatologia, Napoli, Campania
  - UNI DEGLI STUDI - POLICLINICA S. ORSOLA; Dipartimento Malattie dell'Apparato Digerente e Medicina In, Bologna, Emilia-Romagna
  - Az. Osp. Uni Ria Di Parma; Gastro-Enterology, Parma, Emilia-Romagna
  - Fondazione IRCCS Ospedale Maggiore Policlinico; Gastroenterologia, Milan, Lombardy
  - Ospedale Maggiore Policlinico; Iii Divisione Medicina Generale, Milan, Lombardy
  - Uni Di Cagliari; Dept. Di Scienze Mediche, Cagliari, Sardinia
  - Istituto Di Clinica Medica 1 A; Divisione Di Medicina Generale E Gastroenterologia, Palermo, Sicily
  - Ospedale Cisanello - Az. Osp. Pisana; Unità Operativa Di Gastroenterologia Ed Epatologia, Pisa, Tuscany
  - Az. Osp. Di Padova; Dipart. Scienze Chirurgiche E Gastroent., Padua, Veneto
- Auckland Hospital; New Zealand Liver Transplant Unit, Auckland, New Zealand
- Poland (8):
  - Hospital For Infectious Diseases; Infectiology, Bydgoszcz
  - Szpital Specjalistyczny; Oddzial Obserwacyjno - Zakayny, Chorzów
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II; Oddzial Wirusowego Zapalenia Watroby, Krakow
  - Specjalistyczny Szpital Wojewódzki im. Biegańskiego; Klinika Chorób Zakaźnych i Hepatologii UM, Lodz
  - Wojewodzki Szpital Zakazny; Klinika Chorob Zakaznych, Warsaw
  - Centralny Szpital Kliniczny MSWiA; Oddzial Chorob Wewnetrznych i Hepatologii, Warsaw
  - NZOZ Lubuska Specjalistyczna Poradnia Chorob Watroby, Zielona Góra
  - Centrum Medyczne, Łańcut
- Portugal (3):
  - Hospital de Santa Maria; Servico de Gastrenterologia e Hepatologia, Lisbon
  - Hospital Geral de Santo Antonio; Servico de Gastrenterologia, Porto
  - Hospital de Sao Joao; Servico de Gastrenterologia, Porto
- Romania (3):
  - Institutul De Boli Infectioase Matei Bals; Sectia Clinica II Boli Infectioase Adulti, Bucharest
  - The Hospital of Tropical and Infectious Disease Victor Babes, Bucharest
  - Clinical Infectious Diseases Hospital Victor Babes, Craiova
- South Korea (3):
  - Inje University Busan Paik Hospital; Nephrology, Busan
  - Chooncheon Sacred Heart Hospital, Chooncheon
  - Samsung Medical Center; Gastroenterology, Seoul
- Taiwan (9):
  - Changhua Christian Hospital; Internal Medicine, Changhua
  - Kaohsiung Chang Gung Memorial Hospital; Dept of Internal Medicine, Kaohsiung City
  - Kaohsiung Medical Uni Chung-Ho Memorial Hospital; Dept of Internal Medicine, Kaohsiung City
  - Chang Gung Medical Foundation - Keelung; Dept. of Hepato-Gastroenterology, Keelung
  - China Medical University Hospital; Department of Rheumatology, Taichung
  - National Taiwan Uni Hospital; Gastro-Enterology Dept., Taipei
  - Taipei Veterans General Hospital; Gastroenterology Division, Taipei
  - Tri-Service Hospital; Dept. of Internal Medicine, Taipei
  - Chang Gung Medical Foundation - Linkou; Dept. of Hepato-Gastroenterology, Taoyuan District
- Thailand (3):
  - Siriraj Hospital, Bangkok
  - Chiang Mai Uni Hospital; Faculty of Medicine, Chiang Mai
  - Songklanagarind Hospital; Division of Gastroenterology, Songkhla
- United Kingdom (2):
  - The Royal London Hospital, London
  - Manchester Royal Infirmary; Department Of Medicine, Manchester

REFERENCES:
- [Derived] Wei L, Pavlovic V, Bansal AT, Chen X, Foster GR, He H, Kao JH, Lampertico P, Liaw YF, Motoc A, Papatheodoridis GV, Piratvisuth T, Plesniak R, Wat C. Genetic variation in FCER1A predicts peginterferon alfa-2a-induced hepatitis B surface antigen clearance in East Asian patients with chronic hepatitis B. J Viral Hepat. 2019 Sep;26(9):1040-1049. doi: 10.1111/jvh.13107. Epub 2019 Jul 23. PMID 30972912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from Roche completed/ongoing pegylated interferon (Peg-IFN) alfa-2a trials (MV22430/NCT00927082, ML21827/NCT00922207, ML18253/NCT01095835) or from clinical practice (GV28855/NCT01855997).
Groups:
- Adult Participants Treated With Peg-IFN: Adult participants with hepatitis B envelope antigen (HBeAg)-positive or -negative chronic hepatitis B (CHB) infection who completed greater than or equal to (≥) 24 weeks of Peg-IFN alfa-2a (alone or in combination with nucleos[t]ide analogues) therapy and ≥24 weeks of post-treatment follow-up were included. Participants were recruited from Roche clinical trials or general practice; no treatment was administered in this non-interventional study.
Period: Overall Study
Arm/Group | Adult Participants Treated With Peg-IFN
Started | 1669
Completed | 1669
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled Population: All participants for whom genotype data were available.
Groups:
- Adult Participants Treated With Peg-IFN: Adult participants with HBeAg-positive or -negative CHB infection who completed ≥24 weeks of Peg-IFN alfa-2a (alone or in combination with nucleos[t]ide analogues) therapy and ≥24 weeks of post-treatment follow-up were included. Participants were recruited from Roche clinical trials or general practice; no treatment was administered in this non-interventional study.
Arm/Group | Adult Participants Treated With Peg-IFN
Number analyzed (Participants) | 1669
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.09 (0.270)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 471
  Male | 1198
HBeAg Status [Number; unit: participants]
  Positive | 932
  Negative | 676
  Not Known | 61

OUTCOME MEASURES:

1. Primary Outcome: Single Nucleotide Polymorphisms (SNPs) Associated With HBeAg Seroconversion or Hepatitis B Surface Antigen (HBsAg) Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive East Asian (CN) Population: Additive Model
Description: Genome-wide association study (GWAS) approach was used to evaluate the association of SNPs with treatment response. HBeAg seroconversion was defined as the loss of HBeAg and detection of the antibody to HBeAg (anti-HBe). HBsAg clearance was defined as the loss of HBsAg, with or without detection of the antibody to HBsAg (anti-HBs). Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to additive models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive CN Population: All HBeAg-positive participants whose genetic data passed a protocol-specified quality check and shared common East Asian genetic background as compared to haplotype map (HapMap) version 3.0 reference individuals.
Measure: Number; unit: beta coefficient
Groups:
- HBeAg-Positive CN Participants Treated With Peg-IFN: Adult East Asian participants with HBeAg-positive CHB infection who completed ≥24 weeks of Peg-IFN alfa-2a (alone or in combination with nucleos[t]ide analogues) therapy and ≥24 weeks of post-treatment follow-up were included. Participants were recruited from Roche clinical trials or general practice; no treatment was administered in this non-interventional study.
Arm/Group | HBeAg-Positive CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 819
beta coefficient
  rs1876154 | 2.1010
  rs2812338 | 1.8580
  rs10824875 | 1.8330
  rs1831559 | 1.8590
  rs10851257 | 1.8340
  rs6492344 | 1.8120
  rs12584550 | 1.7900
  rs9555773 | 1.8610
  rs7983441 | 1.8770
  rs12446868 | 0.5302
  rs247878 | 0.5209
Statistical Analysis 1: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs1876154; Test type: Superiority or Other; p = 0.00000559, t-test, 2 sided
Statistical Analysis 2: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs2812338; Test type: Superiority or Other; p = 0.00000766, t-test, 2 sided
Statistical Analysis 3: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs10824875; Test type: Superiority or Other; p = 0.00000982, t-test, 2 sided
Statistical Analysis 4: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs1831559; Test type: Superiority or Other; p = 0.00000127, t-test, 2 sided
Statistical Analysis 5: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs10851257; Test type: Superiority or Other; p = 0.00000396, t-test, 2 sided
Statistical Analysis 6: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs6492344; Test type: Superiority or Other; p = 0.00000648, t-test, 2 sided
Statistical Analysis 7: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs12584550; Test type: Superiority or Other; p = 0.00000221, t-test, 2 sided
Statistical Analysis 8: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs9555773; Test type: Superiority or Other; p = 0.00000902, t-test, 2 sided
Statistical Analysis 9: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs7983441; Test type: Superiority or Other; p = 0.00000077, t-test, 2 sided
Statistical Analysis 10: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs12446868; Test type: Superiority or Other; p = 0.00000048, t-test, 2 sided
Statistical Analysis 11: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs247878; Test type: Superiority or Other; p = 0.00000037, t-test, 2 sided

2. Primary Outcome: SNPs Associated With HBeAg Seroconversion or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive CN Population: Dominant Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBeAg seroconversion was defined as the loss of HBeAg and detection of anti-HBe. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to dominant models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive CN Population.
Measure: Number; unit: beta coefficient
Arm/Group | HBeAg-Positive CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 819
beta coefficient
  rs1876154 | 2.2030
  rs7753766 | 2.1200
  rs604241 | 0.4876
  rs12446868 | 0.4501
  rs247878 | 0.4644
Statistical Analysis 1: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs1876154; Test type: Superiority or Other; p = 0.00000987, t-test, 2 sided
Statistical Analysis 2: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs7753766; Test type: Superiority or Other; p = 0.00000605, t-test, 2 sided
Statistical Analysis 3: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs604241; Test type: Superiority or Other; p = 0.00000946, t-test, 2 sided
Statistical Analysis 4: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs12446868; Test type: Superiority or Other; p = 0.00000077, t-test, 2 sided
Statistical Analysis 5: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs247878; Test type: Superiority or Other; p = 0.00000197, t-test, 2 sided

3. Primary Outcome: SNPs Associated With HBeAg Seroconversion or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive Population: Additive Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBeAg seroconversion was defined as the loss of HBeAg and detection of anti-HBe. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to additive models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive Population: All HBeAg-positive participants whose genetic data passed a protocol-specified quality check.
Measure: Number; unit: beta coefficient
Groups:
- HBeAg-Positive Participants Treated With Peg-IFN: Adult participants with HBeAg-positive CHB infection who completed ≥24 weeks of Peg-IFN alfa-2a (alone or in combination with nucleos[t]ide analogues) therapy and ≥24 weeks of post-treatment follow-up were included. Participants were recruited from Roche clinical trials or general practice; no treatment was administered in this non-interventional study.
Arm/Group | HBeAg-Positive Participants Treated With Peg-IFN
Number analyzed (Participants) | 907
beta coefficient
  rs12210761 | 2.7870
  rs1831559 | 1.7250
  rs7983441 | 1.7410
  rs12446868 | 0.5740
  rs247878 | 0.5683
Statistical Analysis 1: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs12210761; Test type: Superiority or Other; p = 0.00000677, t-test, 2 sided
Statistical Analysis 2: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs1831559; Test type: Superiority or Other; p = 0.00000798, t-test, 2 sided
Statistical Analysis 3: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs7983441; Test type: Superiority or Other; p = 0.00000512, t-test, 2 sided
Statistical Analysis 4: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs12446868; Test type: Superiority or Other; p = 0.00000345, t-test, 2 sided
Statistical Analysis 5: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs247878; Test type: Superiority or Other; p = 0.00000372, t-test, 2 sided

4. Primary Outcome: SNPs Associated With HBeAg Seroconversion or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive Population: Dominant Model
Description: as for outcome 2
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive Population.
Measure: Number; unit: beta coefficient
Arm/Group | HBeAg-Positive Participants Treated With Peg-IFN
Number analyzed (Participants) | 907
beta coefficient
  rs12210761 | 3.0040
  rs1411283 | 0.4873
  rs12446868 | 0.5002
Statistical Analysis 1: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs12210761; Test type: Superiority or Other; p = 0.00000459, t-test, 2 sided
Statistical Analysis 2: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs1411283; Test type: Superiority or Other; p = 0.00000925, t-test, 2 sided
Statistical Analysis 3: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs12446868; Test type: Superiority or Other; p = 0.00000772, t-test, 2 sided

5. Primary Outcome: SNPs Associated With HBeAg Seroconversion Plus Undetectable Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive CN Population: Additive Model
Description: GWAS approach was used to evaluate association of SNPs with treatment response. HBeAg seroconversion was defined as the loss of HBeAg and detection of anti-HBe. Undetectable HBV DNA was defined as HBV DNA level below the lower limit of detection (LLD) of 2000 international units per milliliter (IU/mL). HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. HBeAg seroconversion and undetectable HBV DNA were a combined criterion in treatment response. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to additive models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive CN Population.
Measure: Number; unit: beta coefficient
Arm/Group | HBeAg-Positive CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 819
beta coefficient
  rs11163805 | 1.8610
  rs6443144 | 1.9390
  rs11139349 | 1.8360
  rs1831559 | 1.9060
  rs7983441 | 1.9240
  rs11868362 | 0.3363
Statistical Analysis 1: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs11163805; Test type: Superiority or Other; p = 0.00000470, t-test, 2 sided
Statistical Analysis 2: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs6443144; Test type: Superiority or Other; p = 0.00000674, t-test, 2 sided
Statistical Analysis 3: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs11139349; Test type: Superiority or Other; p = 0.00000952, t-test, 2 sided
Statistical Analysis 4: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs1831559; Test type: Superiority or Other; p = 0.00000608, t-test, 2 sided
Statistical Analysis 5: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs7983441; Test type: Superiority or Other; p = 0.00000404, t-test, 2 sided
Statistical Analysis 6: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs11868362; Test type: Superiority or Other; p = 0.00000407, t-test, 2 sided

6. Primary Outcome: SNPs Associated With HBeAg Seroconversion Plus Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive CN Population: Dominant Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBeAg seroconversion was defined as the loss of HBeAg and detection of anti-HBe. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. HBeAg seroconversion and undetectable HBV DNA were a combined criterion in treatment response. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to dominant models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive CN Population.
Measure: Number; unit: beta coefficient
Arm/Group | HBeAg-Positive CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 819
beta coefficient
  rs1384010 | 2.6700
  rs1351518 | 2.3000
  rs1157322 | 3.0120
  rs11868362 | 0.3108
Statistical Analysis 1: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs1384010; Test type: Superiority or Other; p = 0.00000666, t-test, 2 sided
Statistical Analysis 2: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs1351518; Test type: Superiority or Other; p = 0.00000844, t-test, 2 sided
Statistical Analysis 3: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs1157322; Test type: Superiority or Other; p = 0.00000794, t-test, 2 sided
Statistical Analysis 4: Comparison: HBeAg-Positive CN Participants Treated With Peg-IFN; rs11868362; Test type: Superiority or Other; p = 0.00000310, t-test, 2 sided

7. Primary Outcome: SNPs Associated With HBeAg Seroconversion Plus Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive Population: Additive Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBeAg seroconversion was defined as the loss of HBeAg and detection of anti-HBe. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. HBeAg seroconversion and undetectable HBV DNA were a combined criterion in treatment response. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to additive models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive Population.
Measure: Number; unit: beta coefficient
Arm/Group | HBeAg-Positive Participants Treated With Peg-IFN
Number analyzed (Participants) | 907
beta coefficient
  rs11139349 | 1.8610
  rs1157322 | 2.8290
Statistical Analysis 1: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs11139349; Test type: Superiority or Other; p = 0.00000207, t-test, 2 sided
Statistical Analysis 2: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs1157322; Test type: Superiority or Other; p = 0.00000899, t-test, 2 sided

8. Primary Outcome: SNPs Associated With HBeAg Seroconversion Plus Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive Population: Dominant Model
Description: as for outcome 6
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive Population.
Measure: Number; unit: beta coefficient
Arm/Group | HBeAg-Positive Participants Treated With Peg-IFN
Number analyzed (Participants) | 907
beta coefficient
  rs1384010 | 2.6260
  rs1351518 | 2.2220
  rs1157322 | 2.9500
  rs646097 | 0.4639
Statistical Analysis 1: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs1384010; Test type: Superiority or Other; p = 0.00000573, t-test, 2 sided
Statistical Analysis 2: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs1351518; Test type: Superiority or Other; p = 0.00000946, t-test, 2 sided
Statistical Analysis 3: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs1157322; Test type: Superiority or Other; p = 0.00000731, t-test, 2 sided
Statistical Analysis 4: Comparison: HBeAg-Positive Participants Treated With Peg-IFN; rs646097; Test type: Superiority or Other; p = 0.00000945, t-test, 2 sided

9. Primary Outcome: SNPs Associated With Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Negative Non-East Asian (Non-CN) Population: Additive Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to additive models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response. Only a single SNP (rs17037122) was included in the analysis.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Negative Non-CN Population: All HBeAg-negative participants whose genetic data passed a protocol-specified quality check and did not share common East Asian genetic background as compared to HapMap version 3.0 reference individuals.
Measure: Number; unit: beta coefficient
Groups:
- HBeAg-Negative Non-CN Participants Treated With Peg-IFN: Adult non-East Asian participants with HBeAg-negative CHB infection who completed ≥24 weeks of Peg-IFN alfa-2a (alone or in combination with nucleos[t]ide analogues) therapy and ≥24 weeks of post-treatment follow-up were included. Participants were recruited from Roche clinical trials or general practice; no treatment was administered in this non-interventional study.
Arm/Group | HBeAg-Negative Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 371
beta coefficient | 4.3170
Statistical Analysis 1: Comparison: HBeAg-Negative Non-CN Participants Treated With Peg-IFN; rs17037122; Test type: Superiority or Other; p = 0.00000016, t-test, 2 sided

10. Primary Outcome: SNPs Associated With Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Negative Non-CN Population: Dominant Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to dominant models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response. Only a single SNP (rs17037122) was included in the analysis.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Negative Non-CN Population.
Measure: Number; unit: beta coefficient
Arm/Group | HBeAg-Negative Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 371
beta coefficient | 4.2450
Statistical Analysis 1: Comparison: HBeAg-Negative Non-CN Participants Treated With Peg-IFN; rs17037122; Test type: Superiority or Other; p = 0.00000088, t-test, 2 sided

11. Primary Outcome: SNPs Associated With Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Negative CN Population: Additive Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to additive models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response. Only a single SNP (rs2464266) was included in the analysis.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Negative CN Population: All HBeAg-negative participants whose genetic data passed a protocol-specified quality check and shared common East Asian genetic background as compared to HapMap version 3.0 reference individuals.
Measure: Number; unit: beta coefficient
Groups:
- HBeAg-Negative CN Participants Treated With Peg-IFN: Adult East Asian participants with HBeAg-negative CHB infection who completed ≥24 weeks of Peg-IFN alfa-2a (alone or in combination with nucleos[t]ide analogues) therapy and ≥24 weeks of post-treatment follow-up were included. Participants were recruited from Roche clinical trials or general practice; no treatment was administered in this non-interventional study.
Arm/Group | HBeAg-Negative CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 267
beta coefficient | 0.2583
Statistical Analysis 1: Comparison: HBeAg-Negative CN Participants Treated With Peg-IFN; rs2464266; Test type: Superiority or Other; p = 0.00000879, t-test, 2 sided

12. Primary Outcome: SNPs Associated With Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Negative CN Population: Dominant Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to dominant models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Negative CN Population.
Measure: Number; unit: beta coefficient
Arm/Group | HBeAg-Negative CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 267
beta coefficient
  rs9496139 | 0.1812
  rs2014238 | 5.8110
  rs2980231 | 5.8110
Statistical Analysis 1: Comparison: HBeAg-Negative CN Participants Treated With Peg-IFN; rs9496139; Test type: Superiority or Other; p = 0.00000452, t-test, 2 sided
Statistical Analysis 2: Comparison: HBeAg-Negative CN Participants Treated With Peg-IFN; rs2014238; Test type: Superiority or Other; p = 0.00000497, t-test, 2 sided
Statistical Analysis 3: Comparison: HBeAg-Negative CN Participants Treated With Peg-IFN; rs2980231; Test type: Superiority or Other; p = 0.00000497, t-test, 2 sided

13. Primary Outcome: SNPs Associated With Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Negative Population: Additive Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to additive models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Negative Population: All HBeAg-negative participants whose genetic data passed a protocol-specified quality check.
Measure: Number; unit: beta coefficient
Groups:
- HBeAg-Negative Participants Treated With Peg-IFN: Adult participants with HBeAg-negative CHB infection who completed ≥24 weeks of Peg-IFN alfa-2a (alone or in combination with nucleos[t]ide analogues) therapy and ≥24 weeks of post-treatment follow-up were included. Participants were recruited from Roche clinical trials or general practice; no treatment was administered in this non-interventional study.
Arm/Group | HBeAg-Negative Participants Treated With Peg-IFN
Number analyzed (Participants) | 638
beta coefficient
  exm2237722 | 0.1070
  rs16924016 | 0.3357
  rs2899723 | 2.0360
  rs8027115 | 1.9480
  exm2267780 | 2.0100
Statistical Analysis 1: Comparison: HBeAg-Negative Participants Treated With Peg-IFN; exm2237722; Test type: Superiority or Other; p = 0.00000748, t-test, 2 sided
Statistical Analysis 2: Comparison: HBeAg-Negative Participants Treated With Peg-IFN; rs16924016; Test type: Superiority or Other; p = 0.00000073, t-test, 2 sided
Statistical Analysis 3: Comparison: HBeAg-Negative Participants Treated With Peg-IFN; rs2899723; Test type: Superiority or Other; p = 0.00000289, t-test, 2 sided
Statistical Analysis 4: Comparison: HBeAg-Negative Participants Treated With Peg-IFN; rs8027115; Test type: Superiority or Other; p = 0.00000912, t-test, 2 sided
Statistical Analysis 5: Comparison: HBeAg-Negative Participants Treated With Peg-IFN; exm2267780; Test type: Superiority or Other; p = 0.00000494, t-test, 2 sided

14. Primary Outcome: SNPs Associated With Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Negative Population: Dominant Model
Description: as for outcome 12
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Negative Population.
Measure: Number; unit: beta coefficient
Arm/Group | HBeAg-Negative Participants Treated With Peg-IFN
Number analyzed (Participants) | 638
beta coefficient
  rs9973954 | 0.2975
  exm2237722 | 0.1009
  rs1040084 | 2.3660
  rs1913484 | 2.3610
  rs16924016 | 0.3186
  exm1010813 | 0.1299
  rs6576456 | 0.4112
Statistical Analysis 1: Comparison: HBeAg-Negative Participants Treated With Peg-IFN; rs9973954; Test type: Superiority or Other; p = 0.00000627, t-test, 2 sided
Statistical Analysis 2: Comparison: HBeAg-Negative Participants Treated With Peg-IFN; exm2237722; Test type: Superiority or Other; p = 0.00000696, t-test, 2 sided
Statistical Analysis 3: Comparison: HBeAg-Negative Participants Treated With Peg-IFN; rs1040084; Test type: Superiority or Other; p = 0.00000426, t-test, 2 sided
Statistical Analysis 4: Comparison: HBeAg-Negative Participants Treated With Peg-IFN; rs1913484; Test type: Superiority or Other; p = 0.00000435, t-test, 2 sided
Statistical Analysis 5: Comparison: HBeAg-Negative Participants Treated With Peg-IFN; rs16924016; Test type: Superiority or Other; p = 0.00000221, t-test, 2 sided
Statistical Analysis 6: Comparison: HBeAg-Negative Participants Treated With Peg-IFN; exm1010813; Test type: Superiority or Other; p = 0.00000523, t-test, 2 sided
Statistical Analysis 7: Comparison: HBeAg-Negative Participants Treated With Peg-IFN; rs6576456; Test type: Superiority or Other; p = 0.00000757, t-test, 2 sided

15. Primary Outcome: SNPs Associated With HBeAg Seroconversion, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment in Non-CN Population: Additive Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBeAg seroconversion was defined as the loss of HBeAg and detection of anti-HBe. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to additive models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: Non-CN Population: All participants, regardless of HBeAg status, whose genetic data passed a protocol-specified quality check and did not share common East Asian genetic background as compared to HapMap version 3.0 reference individuals.
Measure: Number; unit: beta coefficient
Groups:
- Adult Non-CN Participants Treated With Peg-IFN: Adult non-East Asian participants with HBeAg-positive or -negative CHB infection who completed ≥24 weeks of Peg-IFN alfa-2a (alone or in combination with nucleos[t]ide analogues) therapy and ≥24 weeks of post-treatment follow-up were included. Participants were recruited from Roche clinical trials or general practice; no treatment was administered in this non-interventional study.
Arm/Group | Adult Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 459
beta coefficient
  rs17037122 | 2.9930
  rs10475403 | 0.5024
  rs715243 | 0.5078
Statistical Analysis 1: Comparison: Adult Non-CN Participants Treated With Peg-IFN; rs17037122; Test type: Superiority or Other; p = 0.00000153, t-test, 2 sided
Statistical Analysis 2: Comparison: Adult Non-CN Participants Treated With Peg-IFN; rs10475403; Test type: Superiority or Other; p = 0.00000708, t-test, 2 sided
Statistical Analysis 3: Comparison: Adult Non-CN Participants Treated With Peg-IFN; rs715243; Test type: Superiority or Other; p = 0.00000727, t-test, 2 sided

16. Primary Outcome: SNPs Associated With HBeAg Seroconversion, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment in Non-CN Population: Dominant Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBeAg seroconversion was defined as the loss of HBeAg and detection of anti-HBe. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to dominant models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response. Only a single SNP (rs17037122) was included in the analysis.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: Non-CN Population.
Measure: Number; unit: beta coefficient
Arm/Group | Adult Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 459
beta coefficient | 3.1610
Statistical Analysis 1: Comparison: Adult Non-CN Participants Treated With Peg-IFN; rs17037122; Test type: Superiority or Other; p = 0.00000397, t-test, 2 sided

17. Primary Outcome: SNPs Associated With HBeAg Seroconversion, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment in CN Population: Additive Model
Description: as for outcome 15
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: CN Population: All participants, regardless of HBeAg status, whose genetic data passed a protocol-specified quality check and shared common East Asian genetic background as compared to HapMap version 3.0 reference individuals; the analysis only included a subset of participants who provided evaluable data.
Measure: Number; unit: beta coefficient
Groups:
- Adult CN Participants Treated With Peg-IFN: Adult East Asian participants with HBeAg-positive or -negative CHB infection who completed ≥24 weeks of Peg-IFN alfa-2a (alone or in combination with nucleos[t]ide analogues) therapy and ≥24 weeks of post-treatment follow-up were included. Participants were recruited from Roche clinical trials or general practice; no treatment was administered in this non-interventional study.
Arm/Group | Adult CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 1086
beta coefficient
  rs6443144 | 1.6780
  rs2189452 | 0.6008
  rs9324018 | 1.6680
Statistical Analysis 1: Comparison: Adult CN Participants Treated With Peg-IFN; rs6443144; Test type: Superiority or Other; p = 0.00000686, t-test, 2 sided
Statistical Analysis 2: Comparison: Adult CN Participants Treated With Peg-IFN; rs2189452; Test type: Superiority or Other; p = 0.00000596, t-test, 2 sided
Statistical Analysis 3: Comparison: Adult CN Participants Treated With Peg-IFN; rs9324018; Test type: Superiority or Other; p = 0.00000489, t-test, 2 sided

18. Primary Outcome: SNPs Associated With HBeAg Seroconversion, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment in CN Population: Dominant Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBeAg seroconversion was defined as the loss of HBeAg and detection of anti-HBe. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to dominant models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: CN Population; the analysis only included a subset of participants who provided evaluable data.
Measure: Number; unit: beta coefficient
Arm/Group | Adult CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 1086
beta coefficient
  rs2189452 | 0.5360
  rs7968170 | 0.4869
  rs9324018 | 1.8700
Statistical Analysis 1: Comparison: Adult CN Participants Treated With Peg-IFN; rs2189452; Test type: Superiority or Other; p = 0.00000834, t-test, 2 sided
Statistical Analysis 2: Comparison: Adult CN Participants Treated With Peg-IFN; rs7968170; Test type: Superiority or Other; p = 0.00000487, t-test, 2 sided
Statistical Analysis 3: Comparison: Adult CN Participants Treated With Peg-IFN; rs9324018; Test type: Superiority or Other; p = 0.00000918, t-test, 2 sided

19. Primary Outcome: SNPs Associated With HBeAg Seroconversion, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment: Additive Model
Description: as for outcome 15
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: Genetic Data Quality Check (GT) Population: All participants, regardless of HBeAg status, whose genetic data passed a protocol-specified quality check.
Measure: Number; unit: beta coefficient
Arm/Group | Adult Participants Treated With Peg-IFN
Number analyzed (Participants) | 1545
beta coefficient
  rs9287655 | 0.6617
  rs2803073 | 1.5160
  rs1937590 | 1.7220
  rs2945861 | 0.5957
  rs1997894 | 0.6814
  rs1495471 | 1.5540
  rs9324018 | 1.5400
  rs1152537 | 1.7800
Statistical Analysis 1: Comparison: Adult Participants Treated With Peg-IFN; rs9287655; Test type: Superiority or Other; p = 0.00000137, t-test, 2 sided
Statistical Analysis 2: Comparison: Adult Participants Treated With Peg-IFN; rs2803073; Test type: Superiority or Other; p = 0.00000339, t-test, 2 sided
Statistical Analysis 3: Comparison: Adult Participants Treated With Peg-IFN; rs1937590; Test type: Superiority or Other; p = 0.00000927, t-test, 2 sided
Statistical Analysis 4: Comparison: Adult Participants Treated With Peg-IFN; rs2945861; Test type: Superiority or Other; p = 0.00000166, t-test, 2 sided
Statistical Analysis 5: Comparison: Adult Participants Treated With Peg-IFN; rs1997894; Test type: Superiority or Other; p = 0.00000455, t-test, 2 sided
Statistical Analysis 6: Comparison: Adult Participants Treated With Peg-IFN; rs1495471; Test type: Superiority or Other; p = 0.00000568, t-test, 2 sided
Statistical Analysis 7: Comparison: Adult Participants Treated With Peg-IFN; rs9324018; Test type: Superiority or Other; p = 0.00000125, t-test, 2 sided
Statistical Analysis 8: Comparison: Adult Participants Treated With Peg-IFN; rs1152537; Test type: Superiority or Other; p = 0.00000982, t-test, 2 sided

20. Primary Outcome: SNPs Associated With HBeAg Seroconversion, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment: Dominant Model
Description: as for outcome 18
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: GT Population.
Measure: Number; unit: beta coefficient
Arm/Group | Adult Participants Treated With Peg-IFN
Number analyzed (Participants) | 1545
beta coefficient
  rs10236906 | 0.5664
  rs2945861 | 0.5576
  rs7042473 | 1.7050
  rs2077415 | 0.5732
  rs9324018 | 1.6850
Statistical Analysis 1: Comparison: Adult Participants Treated With Peg-IFN; rs10236906; Test type: Superiority or Other; p = 0.00000846, t-test, 2 sided
Statistical Analysis 2: Comparison: Adult Participants Treated With Peg-IFN; rs2945861; Test type: Superiority or Other; p = 0.00000562, t-test, 2 sided
Statistical Analysis 3: Comparison: Adult Participants Treated With Peg-IFN; rs7042473; Test type: Superiority or Other; p = 0.00000497, t-test, 2 sided
Statistical Analysis 4: Comparison: Adult Participants Treated With Peg-IFN; rs2077415; Test type: Superiority or Other; p = 0.00000997, t-test, 2 sided
Statistical Analysis 5: Comparison: Adult Participants Treated With Peg-IFN; rs9324018; Test type: Superiority or Other; p = 0.00000864, t-test, 2 sided

21. Primary Outcome: SNPs Associated With HBeAg Seroconversion Plus Undetectable HBV DNA, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment in Non-CN Population: Additive Model
Description: as for outcome 7
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: Non-CN Population.
Measure: Number; unit: beta coefficient
Arm/Group | Adult Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 459
beta coefficient
  rs17037122 | 2.8740
  rs715243 | 0.5000
Statistical Analysis 1: Comparison: Adult Non-CN Participants Treated With Peg-IFN; rs17037122; Test type: Superiority or Other; p = 0.00000368, t-test, 2 sided
Statistical Analysis 2: Comparison: Adult Non-CN Participants Treated With Peg-IFN; rs715243; Test type: Superiority or Other; p = 0.00000577, t-test, 2 sided

22. Primary Outcome: SNPs Associated With HBeAg Seroconversion Plus Undetectable HBV DNA, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment in Non-CN Population: Dominant Model
Description: as for outcome 6
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: Non-CN Population.
Measure: Number; unit: beta coefficient
Arm/Group | Adult Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 459
beta coefficient
  rs2302503 | 0.3719
  rs6015181 | 2.6740
Statistical Analysis 1: Comparison: Adult Non-CN Participants Treated With Peg-IFN; rs2302503; Test type: Superiority or Other; p = 0.00000950, t-test, 2 sided
Statistical Analysis 2: Comparison: Adult Non-CN Participants Treated With Peg-IFN; rs6015181; Test type: Superiority or Other; p = 0.00000741, t-test, 2 sided

23. Primary Outcome: SNPs Associated With HBeAg Seroconversion Plus Undetectable HBV DNA, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment in CN Population: Additive Model
Description: as for outcome 7
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: CN Population; the analysis only included a subset of participants who provided evaluable data.
Measure: Number; unit: beta coefficient
Arm/Group | Adult CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 1086
beta coefficient
  rs1550116 | 0.5565
  rs1550115 | 0.5565
  rs2082881 | 0.5565
  exm2265462 | 0.5730
  rs6443144 | 1.8390
  rs1403069 | 0.5769
  rs9691873 | 2.2250
  rs8012912 | 1.6200
  rs11158827 | 1.6200
  rs11870323 | 2.1120
  rs4821558 | 0.6146
Statistical Analysis 1: Comparison: Adult CN Participants Treated With Peg-IFN; rs1550116; Test type: Superiority or Other; p = 0.00000805, t-test, 2 sided
Statistical Analysis 2: Comparison: Adult CN Participants Treated With Peg-IFN; rs1550115; Test type: Superiority or Other; p = 0.00000702, t-test, 2 sided
Statistical Analysis 3: Comparison: Adult CN Participants Treated With Peg-IFN; rs2082881; Test type: Superiority or Other; p = 0.00000702, t-test, 2 sided
Statistical Analysis 4: Comparison: Adult CN Participants Treated With Peg-IFN; exm2265462; Test type: Superiority or Other; p = 0.00000743, t-test, 2 sided
Statistical Analysis 5: Comparison: Adult CN Participants Treated With Peg-IFN; rs6443144; Test type: Superiority or Other; p = 0.00000078, t-test, 2 sided
Statistical Analysis 6: Comparison: Adult CN Participants Treated With Peg-IFN; rs1403069; Test type: Superiority or Other; p = 0.00000894, t-test, 2 sided
Statistical Analysis 7: Comparison: Adult CN Participants Treated With Peg-IFN; rs9691873; Test type: Superiority or Other; p = 0.00000571, t-test, 2 sided
Statistical Analysis 8: Comparison: Adult CN Participants Treated With Peg-IFN; rs8012912; Test type: Superiority or Other; p = 0.00000729, t-test, 2 sided
Statistical Analysis 9: Comparison: Adult CN Participants Treated With Peg-IFN; rs11158827; Test type: Superiority or Other; p = 0.00000828, t-test, 2 sided
Statistical Analysis 10: Comparison: Adult CN Participants Treated With Peg-IFN; rs11870323; Test type: Superiority or Other; p = 0.00000885, t-test, 2 sided
Statistical Analysis 11: Comparison: Adult CN Participants Treated With Peg-IFN; rs4821558; Test type: Superiority or Other; p = 0.00000717, t-test, 2 sided

24. Primary Outcome: SNPs Associated With HBeAg Seroconversion Plus Undetectable HBV DNA, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment in CN Population: Dominant Model
Description: as for outcome 6
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: CN Population; the analysis only included a subset of participants who provided evaluable data.
Measure: Number; unit: beta coefficient
Arm/Group | Adult CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 1086
beta coefficient
  rs6443144 | 1.9800
  rs1692421 | 0.5036
  rs1692423 | 0.5029
  rs9691873 | 2.3190
  rs7968170 | 0.4634
Statistical Analysis 1: Comparison: Adult CN Participants Treated With Peg-IFN; rs6443144; Test type: Superiority or Other; p = 0.00000629, t-test, 2 sided
Statistical Analysis 2: Comparison: Adult CN Participants Treated With Peg-IFN; rs1692421; Test type: Superiority or Other; p = 0.00000579, t-test, 2 sided
Statistical Analysis 3: Comparison: Adult CN Participants Treated With Peg-IFN; rs1692423; Test type: Superiority or Other; p = 0.00000553, t-test, 2 sided
Statistical Analysis 4: Comparison: Adult CN Participants Treated With Peg-IFN; rs9691873; Test type: Superiority or Other; p = 0.00000946, t-test, 2 sided
Statistical Analysis 5: Comparison: Adult CN Participants Treated With Peg-IFN; rs7968170; Test type: Superiority or Other; p = 0.00000450, t-test, 2 sided

25. Primary Outcome: SNPs Associated With HBeAg Seroconversion Plus Undetectable HBV DNA, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment: Additive Model
Description: as for outcome 7
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: GT Population.
Measure: Number; unit: beta coefficient
Arm/Group | Adult Participants Treated With Peg-IFN
Number analyzed (Participants) | 1545
beta coefficient
  rs9287655 | 0.6444
  rs216312 | 0.6621
Statistical Analysis 1: Comparison: Adult Participants Treated With Peg-IFN; rs9287655; Test type: Superiority or Other; p = 0.00000118, t-test, 2 sided
Statistical Analysis 2: Comparison: Adult Participants Treated With Peg-IFN; rs216312; Test type: Superiority or Other; p = 0.00000531, t-test, 2 sided

26. Primary Outcome: SNPs Associated With HBeAg Seroconversion Plus Undetectable HBV DNA, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment: Dominant Model
Description: as for outcome 6
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: GT Population.
Measure: Number; unit: beta coefficient
Arm/Group | Adult Participants Treated With Peg-IFN
Number analyzed (Participants) | 1545
beta coefficient
  rs993147 | 0.5210
  rs10978436 | 1.7610
  rs2370220 | 0.5233
  rs2279519 | 1.7460
Statistical Analysis 1: Comparison: Adult Participants Treated With Peg-IFN; rs993147; Test type: Superiority or Other; p = 0.00000593, t-test, 2 sided
Statistical Analysis 2: Comparison: Adult Participants Treated With Peg-IFN; rs10978436; Test type: Superiority or Other; p = 0.00000997, t-test, 2 sided
Statistical Analysis 3: Comparison: Adult Participants Treated With Peg-IFN; rs2370220; Test type: Superiority or Other; p = 0.00000581, t-test, 2 sided
Statistical Analysis 4: Comparison: Adult Participants Treated With Peg-IFN; rs2279519; Test type: Superiority or Other; p = 0.00000802, t-test, 2 sided

27. Primary Outcome: SNPs Associated With HBsAg Clearance ≥24 Weeks Post-Treatment in Non-CN Population: Additive Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to additive models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response. Only a single SNP (rs12992677) was included in the analysis.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: Non-CN Population; the analysis only included a subset of participants who provided evaluable data.
Measure: Number; unit: beta coefficient
Arm/Group | Adult Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 408
beta coefficient | 5.7670
Statistical Analysis 1: Comparison: Adult Non-CN Participants Treated With Peg-IFN; rs12992677; Test type: Superiority or Other; p = 0.00000558, t-test, 2 sided

28. Primary Outcome: SNPs Associated With HBsAg Clearance ≥24 Weeks Post-Treatment in Non-CN Population: Dominant Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to dominant models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response. Only a single SNP (rs12992677) was included in the analysis.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: Non-CN Population; the analysis only included a subset of participants who provided evaluable data.
Measure: Number; unit: beta coefficient
Arm/Group | Adult Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 408
beta coefficient | 8.6340
Statistical Analysis 1: Comparison: Adult Non-CN Participants Treated With Peg-IFN; rs12992677; Test type: Superiority or Other; p = 0.00000990, t-test, 2 sided

29. Primary Outcome: SNPs Associated With HBsAg Clearance ≥24 Weeks Post-Treatment in CN Population: Additive Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to additive models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response. Only a single SNP (rs7549785) was included in the analysis.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: CN Population.
Measure: Number; unit: beta coefficient
Arm/Group | Adult CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 1095
beta coefficient | 8.2240
Statistical Analysis 1: Comparison: Adult CN Participants Treated With Peg-IFN; rs7549785; Test type: Superiority or Other; p = 0.00000048, t-test, 2 sided

30. Primary Outcome: SNPs Associated With HBsAg Clearance ≥24 Weeks Post-Treatment in CN Population: Dominant Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to dominant models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response. Only a single SNP (rs7549785) was included in the analysis.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: CN Population.
Measure: Number; unit: beta coefficient
Arm/Group | Adult CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 1095
beta coefficient | 8.2240
Statistical Analysis 1: Comparison: Adult CN Participants Treated With Peg-IFN; rs7549785; Test type: Superiority or Other; p = 0.00000048, t-test, 2 sided

31. Primary Outcome: SNPs Associated With HBsAg Clearance ≥24 Weeks Post-Treatment: Additive Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to additive models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: GT Population; the analysis only included a subset of participants who provided evaluable data.
Measure: Number; unit: beta coefficient
Arm/Group | Adult Participants Treated With Peg-IFN
Number analyzed (Participants) | 1503
beta coefficient
  rs10814834 | 0.4571
  rs10491723 | 2.1090
  rs6592052 | 6.6180
  rs16943470 | 2.9650
Statistical Analysis 1: Comparison: Adult Participants Treated With Peg-IFN; rs10814834; Test type: Superiority or Other; p = 0.00000738, t-test, 2 sided
Statistical Analysis 2: Comparison: Adult Participants Treated With Peg-IFN; rs10491723; Test type: Superiority or Other; p = 0.00000451, t-test, 2 sided
Statistical Analysis 3: Comparison: Adult Participants Treated With Peg-IFN; rs6592052; Test type: Superiority or Other; p = 0.00000878, t-test, 2 sided
Statistical Analysis 4: Comparison: Adult Participants Treated With Peg-IFN; rs16943470; Test type: Superiority or Other; p = 0.00000521, t-test, 2 sided

32. Primary Outcome: SNPs Associated With HBsAg Clearance ≥24 Weeks Post-Treatment: Dominant Model
Description: GWAS approach was used to evaluate the association of SNPs with treatment response. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Associations with treatment response were analyzed using logistic regression and adjusted for covariates. Markers were coded according to dominant models of inheritance. Markers surpassing p-value thresholds of p<10^-5 and p<5x10^-8 were considered suggestive and genome-wide significant, respectively. Larger beta coefficients correspond to greater likelihood of treatment response. Only a single SNP (rs6592052) was included in the analysis.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: GT Population; the analysis only included a subset of participants who provided evaluable data.
Measure: Number; unit: beta coefficient
Arm/Group | Adult Participants Treated With Peg-IFN
Number analyzed (Participants) | 1503
beta coefficient | 7.8720
Statistical Analysis 1: Comparison: Adult Participants Treated With Peg-IFN; rs6592052; Test type: Superiority or Other; p = 0.00000720, t-test, 2 sided

33. Other Pre Specified Outcome: Number of Participants With HBeAg Seroconversion or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive Population
Description: Single blood samples were used to analyze HBV serology and genotype data at least 24 weeks post-treatment. HBeAg seroconversion was defined as the loss of HBeAg and detection of anti-HBe. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive Population.
Measure: Number; unit: participants
Arm/Group | HBeAg-Positive Participants Treated With Peg-IFN
Number analyzed (Participants) | 907
participants | 276

34. Other Pre Specified Outcome: Number of Participants With HBeAg Seroconversion or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive CN Population
Description: as for outcome 33
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive CN Population.
Measure: Number; unit: participants
Arm/Group | HBeAg-Positive CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 819
participants | 255

35. Other Pre Specified Outcome: Number of Participants With HBeAg Seroconversion or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive Non-CN Population
Description: as for outcome 33
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive Non-CN Population: All HBeAg-positive participants whose genetic data passed a protocol-specified quality check and did not share common East Asian genetic background as compared to HapMap version 3.0 reference individuals.
Measure: Number; unit: participants
Groups:
- HBeAg-Positive Non-CN Participants Treated With Peg-IFN: Adult non-East Asian participants with HBeAg-positive CHB infection who completed ≥24 weeks of Peg-IFN alfa-2a (alone or in combination with nucleos[t]ide analogues) therapy and ≥24 weeks of post-treatment follow-up were included. Participants were recruited from Roche clinical trials or general practice; no treatment was administered in this non-interventional study.
Arm/Group | HBeAg-Positive Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 88
participants | 21

36. Other Pre Specified Outcome: Number of Participants With HBeAg Seroconversion Plus Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive Population
Description: Single blood samples were used to analyze HBV serology and genotype data at least 24 weeks post-treatment. HBeAg seroconversion was defined as the loss of HBeAg and detection of anti-HBe. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. HBeAg seroconversion and undetectable HBV DNA were a combined endpoint in this outcome measure.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive Population.
Measure: Number; unit: participants
Arm/Group | HBeAg-Positive Participants Treated With Peg-IFN
Number analyzed (Participants) | 907
participants | 193

37. Other Pre Specified Outcome: Number of Participants With HBeAg Seroconversion Plus Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive CN Population
Description: as for outcome 36
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive CN Population.
Measure: Number; unit: participants
Arm/Group | HBeAg-Positive CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 819
participants | 175

38. Other Pre Specified Outcome: Number of Participants With HBeAg Seroconversion Plus Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Positive Non-CN Population
Description: as for outcome 36
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Positive Non-CN Population.
Measure: Number; unit: participants
Arm/Group | HBeAg-Positive Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 88
participants | 18

39. Other Pre Specified Outcome: Number of Participants With Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Negative Population
Description: Single blood samples were used to analyze HBV serology and genotype data at least 24 weeks post-treatment. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Negative Population.
Measure: Number; unit: participants
Arm/Group | HBeAg-Negative Participants Treated With Peg-IFN
Number analyzed (Participants) | 638
participants | 393

40. Other Pre Specified Outcome: Number of Participants With Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Negative CN Population
Description: as for outcome 39
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Negative CN Population.
Measure: Number; unit: participants
Arm/Group | HBeAg-Negative CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 267
participants | 209

41. Other Pre Specified Outcome: Number of Participants With Undetectable HBV DNA or HBsAg Clearance ≥24 Weeks Post-Treatment in HBeAg-Negative Non-CN Population
Description: as for outcome 39
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: HBeAg-Negative Non-CN Population.
Measure: Number; unit: participants
Arm/Group | HBeAg-Negative Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 371
participants | 184

42. Other Pre Specified Outcome: Number of Participants With HBeAg Seroconversion, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment
Description: Single blood samples were used to analyze HBV serology and genotype data at least 24 weeks post-treatment. HBeAg seroconversion was defined as the loss of HBeAg and detection of anti-HBe. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs. Undetectable HBV DNA was defined as an HBV DNA level below the LLD of 2000 IU/mL.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: GT Population.
Measure: Number; unit: participants
Arm/Group | Adult Participants Treated With Peg-IFN
Number analyzed (Participants) | 1545
participants | 669

43. Other Pre Specified Outcome: Number of Participants With HBeAg Seroconversion, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment in CN Population
Description: as for outcome 42
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: CN Population; the analysis only included a subset of participants who provided evaluable data.
Measure: Number; unit: participants
Arm/Group | Adult CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 1086
participants | 464

44. Other Pre Specified Outcome: Number of Participants With HBeAg Seroconversion, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment in Non-CN Population
Description: as for outcome 42
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: Non-CN Population.
Measure: Number; unit: participants
Arm/Group | Adult Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 459
participants | 205

45. Other Pre Specified Outcome: Number of Participants With HBeAg Seroconversion Plus Undetectable HBV DNA, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment
Description: as for outcome 36
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: GT Population.
Measure: Number; unit: participants
Arm/Group | Adult Participants Treated With Peg-IFN
Number analyzed (Participants) | 1545
participants | 586

46. Other Pre Specified Outcome: Number of Participants With HBeAg Seroconversion Plus Undetectable HBV DNA, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment in CN Population
Description: as for outcome 36
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: CN Population.
Measure: Number; unit: participants
Arm/Group | Adult CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 1086
participants | 384

47. Other Pre Specified Outcome: Number of Participants With HBeAg Seroconversion Plus Undetectable HBV DNA, HBsAg Clearance, or Undetectable HBV DNA ≥24 Weeks Post-Treatment in Non-CN Population
Description: as for outcome 36
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: Non-CN Population.
Measure: Number; unit: participants
Arm/Group | Adult Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 459
participants | 202

48. Other Pre Specified Outcome: Number of Participants With HBsAg Clearance ≥24 Weeks Post-Treatment
Description: Single blood samples were used to analyze HBV serology and genotype data at least 24 weeks post-treatment. HBsAg clearance was defined as the loss of HBsAg, with or without detection of anti-HBs.
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: GT Population; the analysis only included a subset of participants who provided evaluable data.
Measure: Number; unit: participants
Arm/Group | Adult Participants Treated With Peg-IFN
Number analyzed (Participants) | 1503
participants | 104

49. Other Pre Specified Outcome: Number of Participants With HBsAg Clearance ≥24 Weeks Post-Treatment in CN Population
Description: as for outcome 48
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: CN Population.
Measure: Number; unit: participants
Arm/Group | Adult CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 1095
participants | 80

50. Other Pre Specified Outcome: Number of Participants With HBsAg Clearance ≥24 Weeks Post-Treatment in Non-CN Population
Description: as for outcome 48
Time Frame: Single blood sample ≥24 weeks post-treatment
Population: Non-CN Population; the analysis only included a subset of participants who provided evaluable data.
Measure: Number; unit: participants
Arm/Group | Adult Non-CN Participants Treated With Peg-IFN
Number analyzed (Participants) | 408
participants | 24

ADVERSE EVENTS:
Time Frame: Single visit at least 24 weeks after completion of treatment (overall sampling period up to 12 months)
Description: Participants who were recruited directly into the study from general practice and who provided a blood sample were observed only for adverse events (AEs) related to the blood sampling procedure.
Groups:
- Adult Participants Treated With Peg-IFN: Adult participants with HBeAg-positive or -negative CHB infection, and who had completed at least 24 weeks of Peg-IFN alfa-2a with/without nucleoside analogue therapy and at least 24 weeks of follow-up, were included. Participants were recruited from Roche clinical trials or general practice; no treatment was administered in this non-interventional study.
Arm/Group | Adult Participants Treated With Peg-IFN
Serious Adverse Events (participants affected / at risk) | 0/1105
Other Adverse Events (participants affected / at risk) | 0/1105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.